CLINICAL TRIAL: NCT03267784
Title: An Interventional, Multicenter, Single Arm, Phase I/IIa Clinical Trial to Investigate the Efficacy and Safety of Allo-APZ2-DFU on Wound Healing of Diabetic Neuropathic Ulcer (DFU)
Brief Title: Allogeneic ABCB5-positive Stem Cells for Treatment of DFU "Malum Perforans"
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: RHEACELL GmbH & Co. KG (Industry)
Collaborators: FGK Clinical Research GmbH (Industry); Ticeba GmbH (Industry); Granzer Regulatory Consulting & Services (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: allo-APZ2-DFU-II-01
Record Dates: First submitted 2017-08-17; First posted 2017-08-30 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Diabetic Neuropathic Ulcer
Keywords: diabetic neuropathic ulcer; ABCB5; allogeneic; mesenchymal stem cells; skin ulcer; advanced therapy medicinal product; somatic cell therapy; phase I/IIa; Diabetic Foot Ulcer
MeSH Terms: conditions — Skin Ulcer; Diabetic Foot

STUDY DESIGN:
Intervention Model Description: Single Group Assignment Interventional, single arm, multicenter, phase I/IIa clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: allo-APZ2-DFU (Experimental): Application of IMP on patients wound
  Interventions: Biological: allo-APZ2-DFU

INTERVENTIONS:
Biological: allo-APZ2-DFU — Suspension of ABCB5-positive mesenchymal stem cells

SUMMARY:
The aim of this clinical trial is to investigate the efficacy (by monitoring the wound surface area reduction of Diabetic Foot Ulcers) and safety (by monitoring adverse events) of two doses of the allogeneic investigational medicinal product "allo-APZ2-DFU" topically administered to the wound matrix of patients with diabetic neuropathic ulcer.

DETAILED DESCRIPTION:
This is an interventional, single arm, phase I/IIa clinical trial to investigate the efficacy and safety of allogeneic ABCB5-positive mesenchymal stem cells (MSCs) on wound healing in patients with diabetic neuropathic ulcer. Allogeneic MSCs will be isolated ex vivo and will be expanded in vitro. The Investigational medicinal product (IMP) containing the ABCB5-positive MSCs will then be applied two times (at Visit 3 and six weeks later, at Visit 10) on the wound surface of DFU.

Patients are followed up for efficacy for a period of three months starting after the first IMP application which allows to distinguish actual wound healing from transient wound coverage.

The wound healing process will be documented by standardized photography. The wound size reduction evaluation will start two weeks after the first IMP application. The quality of the wound healing process will be assessed on the basis of formation of granulation tissue, epithelialization and wound exudation.

Pain will be assessed using a numerical rating scale and quality of life will be investigated with standardized and validated questionnaires. To assess long-term safety of allo-APZ2-DFU three follow-up visits at Months 6, 9 and 12 after the first IMP application are included.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged 18 to 85 years;
2. Patients with an existing diagnosis of diabetic mellitus Type 2, evaluated by blood test [HbA1c] < 11%) at the Screening visit (Visit 1). The HbA1c value at visit 1 should not vary more than 1.5% (absolute range) compared to a HbA1c value that was previously measured 1 to 6 months before visit 1;
3. The presence of diabetic neuropathic ulcers "malum perforans" (Grade I and II according to Wagner) at plantar site of the foot diagnosed by ABI ≥0.7, without claudication, or TcPO2 >40 mmHg or doppler ultrasonography (at the discretion of the investigator) to exclude significant arterial diseases and critical limb ischemia, and a diabetic neuropathy test using a 128 Hz vibration tuning fork according to Rydel-Seiffer (as described by Guideline "Nationale Versorgungsleitlinie - Neuropathie bei Diabetes im Erwachsenenalter"). If the ABI is >1.3, an additional doppler ultrasonography must be performed to exclude a PAOD masked by media sclerosis;
4. At Screening Visit 1 and 2 the wound surface area of the target ulcer should be between 1 and 50 cm2 measured by using a scaled measuring sensor in combination with digital image analysis;
5. The ulcer's surface area should be (mostly) free from callus or necrotic tissue;
6. If patients are suffering from two or more ulcers at the same extremity, the target ulcer has to be separated by a minimum bridge of 1 cm of healthy tissue from other ulcers;
7. Patients are willing and able to wear therapeutic shoes that are especially designed for patients with a diabetic neuropathic foot;
8. Body mass index (BMI) between 20 and 45 kg/m²;
9. Patients understand the nature of the procedure and are providing written informed consent prior to any clinical trial procedure;
10. Women of childbearing potential must have a negative blood pregnancy test at Visit 1;
11. Women of childbearing potential must be willing to use highly effective contraceptive methods during the course of the clinical trial.

Exclusion Criteria:

1. Presence of acute Charcot foot;
2. Clinical signs of active osteomyelitis in the last three months;
3. Active wet gangrenous tissue;
4. Infection of the target ulcer requiring treatment as judged clinically;
5. Presence of an ulcer Grade ≥3 according to Wagner on the same foot as target ulcer;
6. Patients who are currently receiving dialysis;
7. Peripheral arterial occlusive disease (PAOD) including claudication with need of treatment;
8. Ulcers due to non-diabetic etiology;
9. Prior surgical procedures such as bypass or mesh-graft treatment within 2 months prior to IMP application;
10. Acute deep vein thrombosis (maximum 30 days from diagnosis) or a still untreated deep vein thrombosis;
11. Any chronic dermatological disorders diagnosed at the investigator's discretion;
12. Skin disorders, unrelated to the ulcer, that are present adjacent to the target wound;
13. Treatment of target wound with active wound care agents (e.g. iruxol, local antibiotics or silver dressings), which have not been stopped 14 days before IMP application;
14. Any malignancy within the past 5 years, excluding successfully treated carcinoma in situ, basal cell carcinoma or squamous cell carcinoma of the skin without evidence of metastases;
15. Current use of steroid medication above Cushing threshold dose (>7.5 mg/d prednisone or equivalent);
16. Known abuse of alcohol, drugs, or medicinal products;
17. Patients anticipated to be unwilling or unable to comply with the requirements of the protocol;
18. Pregnant or lactating women;
19. Patients infected with the human immunodeficiency virus (HIV 1&2);
20. Any known allergies to components of the IMP or concomitant medication;
21. Current or previous (within 30 days of enrollment) treatment with another IMP, or participation and/or under follow-up in another clinical trial;
22. Evidence of any other medical conditions (such as psychiatric illness, physical examination, or laboratory findings) that may interfere with the planned treatment, affect the patient's compliance, or place the patient at high risk of complications related to the treatment;
23. Employees of the sponsor, or employees or relatives of the investigator.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2020-06-29 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Percentage of wound surface area reduction | Week 12, or last available post-baseline measurement of weeks 4, 6 or 8 if the Week 12 measurement is missing.
  Percentage of wound surface area reduction at Week 12, or last available post-baseline measurement of weeks 4, 6 or 8, if the Week 12 measurement is missing (last observation carried forward [LOCF]).
Assessment of adverse event (AE) occurrence | Up to 12 months
  All AEs occurring during the clinical trial will be registered, documented and evaluated.

SECONDARY OUTCOMES:
Percentage of wound surface area reduction | Weeks 2, 4, 6, 8 and 12 (without LOCF)
  Percentage of wound surface area reduction will be evaluated.
Percentage of invisible and visible wound surface area reduction | Weeks 2, 4, 6, 8 and 12 (without LOCF)
  Percentage of invisible and visible wound surface area reduction will be evaluated.
Absolute wound surface area reduction | Weeks 2, 4, 6, 8 and 12 (without LOCF)
  Absolute wound surface area reduction will be evaluated.
Absolute invisible and visible wound surface area reduction | Weeks 2, 4, 6, 8 and 12 (without LOCF)
  Absolute invisible and visible wound surface area reduction will be evaluated.
Assessment of wound infection | Days 1 and 2, Weeks 1, 2, 4, 6, 6.1, 6.2, 6.3, 8 and 12
  Wound infection will be evaluated.
Time to first complete wound closure | A priori specification not possible; between baseline and week 12 post baseline
  Time to first complete wound closure will be evaluated.
Proportion of patients achieving complete wound closure | Weeks 2, 4, 6, 8 and 12
  Proportion of patients achieving complete wound closure will be evaluated.
Time to first 30% reduction of wound surface area | A priori specification not possible; between baseline and week 12 post baseline
  Time to first 30% reduction of wound surface area will be evaluated.
Proportion of patients achieving 30% reduction of wound surface area | Weeks 2, 4, 6, 8 and 12
  Proportion of patients achieving 30% reduction of wound surface area will be evaluated.
Assessment of wound exudation, epithelialization and formation of granulation tissue | Day 0 and Week 6.1 prior IMP-application, at Weeks 1, 2, 4, 6, 8 and 12
  Wound exudation, epithelialization and formation of granulation tissue will be evaluated.
Time to amputation at target leg until Week 12 | A priori specification not possible; between baseline and week 12 post baseline
  Time to amputation at target leg until week 12 will be evaluated.
Pain assessment as per numerical rating scale (NRS) | At both Screening Visits, at Days 0, 1 and 2 and at Weeks 1, 2, 4, 6, 6.1, 6.2, 6.3, 8 and 12
  Pain assessment as per numerical rating scale (NRS) will be evaluated.
Assessment of Quality of life (QoL) using the short form 36 (SF-36) questionnaire | Screening Visit 1, Visit 3, at Weeks 4 and 12
  Quality of life (QoL) using the short form 36 (SF-36) questionnaire will be evaluated.
Assessment of Dermatology-specific QoL based on the Dermatology Life Quality Index (DLQI) questionnaire | Screening Visit 1, Visit 3, at Weeks 4 and 12
  Dermatology-specific QoL based on the Dermatology Life Quality Index (DLQI) questionnaire will be evaluated.
Physical examination and vital signs | Week 6.1 and Week 12
  Physical examination and vital signs will be evaluated.
Time to amputation of target leg until month 12 | A priori specification not possible; between baseline and month 12 post baseline
  Time to amputation of target leg until month 12 will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kerstan, Dr., Principal Investigator — Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Würzburg, Germany
Locations (7):
- Germany (7):
  - Universitätsmedizin Greifswald; Klinik und Poliklinik für Hautkrankheiten, Greifswald
  - St. Josefskrankenhaus Heidelberg GmbH; Klinische Studienabteilung, Heidelberg
  - Diabetologikum Raab, Privatärztliche Facharztpraxis, Kassel
  - pro scientia med im Mare Klinikum, Department Klinische Forschung und Entwicklung, Kronshagen
  - Studienambulanz Leipzig, medamed GmbH, Leipzig
  - Diabetologikum Ludwigshafen, Gemeinschaftspraxis, Ludwigshafen
  - Klinik und Poliklinik für Dermatologie, Venerologie und Allergologie, Universitätsklinikum Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerstan A, Dieter K, Niebergall-Roth E, Klingele S, Junger M, Hasslacher C, Daeschlein G, Stemler L, Meyer-Pannwitt U, Schubert K, Klausmann G, Raab T, Goebeler M, Kraft K, Esterlechner J, Schroder HM, Sadeghi S, Ballikaya S, Gasser M, Waaga-Gasser AM, Murphy GF, Orgill DP, Frank NY, Ganss C, Scharffetter-Kochanek K, Frank MH, Kluth MA. Translational development of ABCB5+ dermal mesenchymal stem cells for therapeutic induction of angiogenesis in non-healing diabetic foot ulcers. Stem Cell Res Ther. 2022 Sep 5;13(1):455. doi: 10.1186/s13287-022-03156-9. PMID 36064604
- [Derived] Kerstan A, Niebergall-Roth E, Esterlechner J, Schroder HM, Gasser M, Waaga-Gasser AM, Goebeler M, Rak K, Schrufer P, Endres S, Hagenbusch P, Kraft K, Dieter K, Ballikaya S, Stemler N, Sadeghi S, Tappenbeck N, Murphy GF, Orgill DP, Frank NY, Ganss C, Scharffetter-Kochanek K, Frank MH, Kluth MA. Ex vivo-expanded highly pure ABCB5+ mesenchymal stromal cells as Good Manufacturing Practice-compliant autologous advanced therapy medicinal product for clinical use: process validation and first in-human data. Cytotherapy. 2021 Feb;23(2):165-175. doi: 10.1016/j.jcyt.2020.08.012. Epub 2020 Oct 1. PMID 33011075